CLINICAL TRIAL: NCT05148156
Title: Reduction of Urinary Toxicity of Stereotactic Body Radiation Therapy (SBRT) With Prostatic Urethral Lift (Urolift)
Brief Title: Urolift Pre-SBRT for Reduced Urinary Toxicity in Patients With BPH and Prostate Cancer.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator changing locations.
Sponsor: Northwell Health (Other)
Collaborators: NeoTract, Inc. (Industry); Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0684
Record Dates: First submitted 2021-11-23; First posted 2021-12-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: stereotactic body radiation therapy; urolift; prostatic urethral lift; dysuria; nocturia; minimally invasive therapy
MeSH Terms: conditions — Prostatic Hyperplasia; Dysuria; Nocturia

STUDY DESIGN:
Intervention Model Description: This is a single-arm study, involving one time administration of Urolift in outpatient setting prior to stereotactic body radiation therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Urolift (Experimental): This is a single-arm study involving 1 year of follow-up. Study intervention involves a one-time administration of Urolift prior to SBRT for prostate cancer treatment.
  Interventions: Device: Urolift

INTERVENTIONS:
Device: Urolift — Study intervention involves a one-time administration of Urolift in out-patient setting prior to Stereotactic body radiation therapy (SBRT).

SUMMARY:
Many patients may face long-term urinary side effects following stereotactic body radiation therapy (SBRT), including increased urinary frequency, dysuria, and nocturia. The investigator hypothesizes that Urolift, which represents a novel minimally invasive therapy, may reduce acute and long-term urinary toxicity and side effects of radiation therapy (SBRT).

DETAILED DESCRIPTION:
Urolift is a standard of care treatment for BPH. It involves the placement of a stainless-steel urethral end piece tethered to a capsular tab to the left and right side of the prostatic urethra approximately 1.5cm distal to the bladder neck. It pulls and maintains the opening of a continuous channel through the prostatic urethra. A previous study examined the effect of Urolift on urinary symptoms and urinary medications at six months post-procedure.Urolift was associated with significant urinary improvements measured by IPSS and quality of life questionnaires and a reduction in the use of total medication as well as alpha-blockers and beta-3 agonists.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 50 - 99 years of age
* Subject has provided informed consent
* Subject has diagnosis of prostate cancer requiring SBRT
* Subject is able to complete self-administered questionnaires
* Subject is a surgical candidate for Urolift
* Subject has a diagnosis of BPH
* Medical record documentation of prostate volume from 30-80 ml by TRUS
* Absence of a middle lobe

Exclusion Criteria:

* Life expectancy < 2 years
* Currently enrolled in or plans to enroll in any concurrent drug or device study
* Concurrent androgen deprivation therapy
* Has an active infection (e.g., urinary tract infection or prostatitis)
* Diagnosis of or has received treatment for chronic prostatitis or chronic pelvic pain syndrome (e.g., nonbacterial chronic prostatitis)
* Subject has been diagnosed with a urethral stricture or bladder neck contracture within the last 180 days
* Subject has been diagnosed with 2 or more urethral strictures and/or bladder neck contractures within 5 years
* Diagnosis of lichen sclerosis
* Neurogenic bladder or other neurologic disorder that affects bladder function
* Diagnosis of polyneuropathy (e.g., diabetic)
* History of lower urinary tract surgery
* Subject has diagnosis of stress urinary incontinence that requires treatment or daily pad or device use
* Subject has been catheterized or has a PVR > 400 ml in the 14 days prior to the surgical procedure
* Current diagnosis of bladder stones

Ages: 50 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in IPSS scores from baseline and one year post treatment | At baseline and one year post treatment
  Patients will take a International Prostatic Symptom Score (IPSS) questionnaire to evaluate symptom severity at baseline and 1 year post treatment. IPSS scores range from 1 to 35, with 1-7 indicating mild symptoms, 8-19 indicating moderate symptoms, 20-35 indicating severe symptoms.
Change in IIEF score through study completion, an average of 1 year | Through study completion, an average of 1 year
  Patient will take the International Index of Erectile Function (IIEF) to evaluate changes in sexual function of patients through study completion, an average of 1 year. IIEF scores range from 6 to 30. IIEF lower scores indicate severe erectile dysfunction, while higher scores indicate mild/no erectile dysfunction.
Change in MSHQ through study completion, an average of 1 year | Through study completion, an average of 1 year
  Patients will take the Men's sexual health questionnaire (MSHQ) to further evaluate patients' ability to have sex with their partner(s) or masturbate through study completion, an average of 1 year.
  Overall, study subjects will be assessed for possible change in hypogonadal, sexual function, and pain symptoms. Scores range from 16 to 125. Lower scores are considered most symptomatic, higher scores are least symptomatic.
Change in VAS score through study completion, an average of 1 year | through study completion, an average of 1 year
  Patients will use a visual analog scale (VAS) to describe their pain through study completion, an average of 1 year, to see if there is any changes in pain post treatment. Self-assessed maximum pain reported using a 0-100mm visual analog scale, where 100 signifies maximum pain and 0 signifies no pain.
Change in OAB-SF score through study completion, an average of 1 year | Through study completion, an average of 1 year
  Patients will use a overactive bladder short form (OAB-SF) to describe their overactive bladder symptoms through study completion, an average of 1 year, to see if there is any changes in symptoms.
  The OAB-q SF has 2 main subscales: Symptom bother and Health-Related Quality of Life (HRQOL). The two subscales are summed separately and transformed into scores ranging from 0 to 100. A higher score on the symptom bother scale indicates a greater symptom severity and a higher score on the HRQOL scale indicates a better HRQOL, so they are inversely related to each other. Since the OAB-q SF has no total score, higher scores indicate more severe symptoms or better quality of life, respectively. Lower scores indicate less severe symptoms or worse quality of life respectively.
Change in SF-12 score through study completion, an average of 1 year | Through study completion, an average of 1 year
  Patients will use a short form 12 (SF-12) survey to measure their quality of life through study completion, an average of 1 year, to see if there is any changes.
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less on the PCS-12 has been recommended as a cut-off to determine a physical condition; while a score of 42 or less on the MCS-12 may be indicative of 'clinical depression'.

SECONDARY OUTCOMES:
Change in medication usage through study completion, an average of 1 year | Through study completion, an average of 1 year
  Patients will list their medication usage through study completion, an average of 1 year to see if there is any changes in medications after the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Syosset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng M, Leslie SW, Baradhi KM. Benign Prostatic Hyperplasia. 2024 Oct 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558920/ PMID 32644346
- [Background] McVary KT. BPH: epidemiology and comorbidities. Am J Manag Care. 2006 Apr;12(5 Suppl):S122-8. PMID 16613526
- [Background] Alcaraz A, Hammerer P, Tubaro A, Schroder FH, Castro R. Is there evidence of a relationship between benign prostatic hyperplasia and prostate cancer? Findings of a literature review. Eur Urol. 2009 Apr;55(4):864-73. doi: 10.1016/j.eururo.2008.11.011. Epub 2008 Nov 21. PMID 19027219
- [Background] Roehrborn CG. Prostatic Urethral Lift: A Unique Minimally Invasive Surgical Treatment of Male Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. Urol Clin North Am. 2016 Aug;43(3):357-69. doi: 10.1016/j.ucl.2016.04.008. PMID 27476128
- [Background] Chialastri P, Chialastri A, Mueller T. Does Prostatic Urethral Lift Reduce Urinary Medications? Trends in Medical Treatment Before and After Prostatic Urethral Lift. J Endourol. 2021 May;35(5):657-662. doi: 10.1089/end.2020.0848. Epub 2021 Jan 20. PMID 33198488
- [Background] Cihan Y. The role and importance of SBRT in prostate cancer. Int Braz J Urol. 2018 Nov-Dec;44(6):1272-1274. doi: 10.1590/S1677-5538.IBJU.2018.0484. No abstract available. PMID 30325604
- [Background] Janowski E, Chen LN, Kim JS, Lei S, Suy S, Collins B, Lynch J, Dritschilo A, Collins S. Stereotactic body radiation therapy (SBRT) for prostate cancer in men with large prostates (>/=50 cm(3)). Radiat Oncol. 2014 Nov 15;9:241. doi: 10.1186/s13014-014-0241-3. PMID 25398516
- [Background] Mbeutcha A, Chauveinc L, Bondiau PY, Chand ME, Durand M, Chevallier D, Amiel J, Kee DL, Hannoun-Levi JM. Salvage prostate re-irradiation using high-dose-rate brachytherapy or focal stereotactic body radiotherapy for local recurrence after definitive radiation therapy. Radiat Oncol. 2017 Mar 9;12(1):49. doi: 10.1186/s13014-017-0789-9. PMID 28274241
- [Background] Fuller DB, Wurzer J, Shirazi R, Bridge SS, Law J, Mardirossian G. High-dose-rate stereotactic body radiation therapy for postradiation therapy locally recurrent prostatic carcinoma: Preliminary prostate-specific antigen response, disease-free survival, and toxicity assessment. Pract Radiat Oncol. 2015 Nov-Dec;5(6):e615-23. doi: 10.1016/j.prro.2015.04.009. Epub 2015 Jun 6. PMID 26059509
- [Background] Jiang P, Krockenberger K, Vonthein R, Tereszczuk J, Schreiber A, Liebau S, Huttenlocher S, Imhoff D, Balermpas P, Keller C, Dellas K, Baumann R, Rodel C, Hildebrandt G, Junemann KP, Merseburger AS, Katz A, Ziegler A, Blanck O, Dunst J. Hypo-fractionated SBRT for localized prostate cancer: a German bi-center single treatment group feasibility trial. Radiat Oncol. 2017 Aug 18;12(1):138. doi: 10.1186/s13014-017-0872-2. PMID 28821268